CLINICAL TRIAL: NCT06233825
Title: Nutritional Intervention to Enhance Recovery After Arthroscopic Knee Surgery in Adults: A Randomized Controlled Pilot Trial
Brief Title: Nutritional Intervention to Enhance Recovery After Arthroscopic Knee Surgery in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Chris McGlory, PhD (Other)
Responsible Party: Sponsor-Investigator, Dr. Chris McGlory, PhD, Assistant Professor, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 6038901
Record Dates: First submitted 2024-01-19; First posted 2024-01-31 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-08

CONDITIONS: Anterior Cruciate Ligament Reconstruction; Muscular Atrophy
Keywords: omega-3 fatty acids; fish oil; eicosapentaenoic acid; docosahexaenoic acid; skeletal muscle; anterior cruciate ligament; essential amino acids; magnetic resonance imaging; muscle protein synthesis
MeSH Terms: conditions — Muscular Atrophy | interventions — Fatty Acids, Omega-3; Amino Acids, Essential; Fish Oils; Safflower Oil

STUDY DESIGN:
Intervention Model Description: Randomized controlled feasibility pilot trial.Two-arm study. Half of participants are allocated to the nutritional intervention condition (5 g omega-3, 40 g essential amino acids [EAA] per day), and half to the placebo control condition (5 g safflower oil, 40 g non-essential amino acids [NEAA] per day).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutritional Intervention (Experimental): 5 g omega-3 fatty acids (3.75 g eicosapentaenoic acid [EPA] + 1.25 g docosahexaenoic acid [DHA]) per day for 6 weeks, starting 4 weeks before and continuing 2 weeks after surgery, plus 40 g (2 x 20 g) of EAA per day, starting 1 week before and continuing 2 weeks after surgery.
  Interventions: Dietary Supplement: Omega-3 Fatty Acids and Essential Amino Acids
- Placebo Control (Placebo Comparator): 5 g safflower oil per day for 6 weeks, starting 4 weeks before and continuing 2 weeks after surgery, plus 40 g (2 x 20 g) of NEAA per day, starting 1 week before and continuing 2 weeks after surgery.
  Interventions: Dietary Supplement: Safflower Oil and Non-Essential Amino Acids

INTERVENTIONS:
Dietary Supplement: Omega-3 Fatty Acids and Essential Amino Acids — Oil consumed as capsules. EAA come as powder to be mixed with water before drinking. 4 g of leucine per EAA dose.
  Other Names: Fish Oil
  Arms: Nutritional Intervention
Dietary Supplement: Safflower Oil and Non-Essential Amino Acids — Oil consumed as capsules. NEAA are isonitrogenous to intervention condition. Both supplement types are isoenergetic to intervention. NEAA come as powder to be mixed with water before drinking.
  Arms: Placebo Control

SUMMARY:
Loss of skeletal muscle mass (atrophy) and strength in the lower limb are consequences of elective knee surgery as result of prolonged disuse from limb immobilization and impaired mobility, as well as pathophysiological trauma. The highest rates of skeletal muscle mass and strength loss occur during the 2-week post-surgery period, considered the early phase of outpatient recovery. Alternative to resistance exercise and pharmacology, nutritional intervention represents one strategy to combat skeletal muscle disuse atrophy.

Essential amino acids (EAA) and omega-3 fatty acids are known to independently potentiate rates of skeletal muscle protein synthesis and attenuate skeletal muscle atrophy in humans. However, the combined actions these nutritional strategies on skeletal muscle have not been explored in a pathophysiological context, such as surgery. With the ultimate goal to test the efficacy of the combined nutritional strategy to attenuate skeletal muscle disuse atrophy in the future, the aim of this present pilot study is to explore the feasibility of recruitment and retention of anterior cruciate ligament reconstruction (ACLR) outpatients from a single centre across 18 months for a 6-week nutritional intervention. Participants will consume either an intervention of omega-3 fatty acids and EAAs, or a placebo control of safflower oil and non-essential amino acids (NEAA), for 4 weeks before and 2 weeks after elective ACLR surgery. Furthermore, this pilot will characterize secondary outcomes of skeletal muscle mass, strength, and power, and integrated rates of muscle protein synthesis, as well as report participant adherence to protocols and incidence of adverse events.

DETAILED DESCRIPTION:
Over their lifespan, many individuals experience episodes of skeletal muscle-disuse due to illness, injury, or elective surgery. Periods of prolonged skeletal muscle disuse, such after ACLR, result in the loss of skeletal muscle mass (atrophy) and strength. Skeletal muscle disuse precipitates several metabolic and functional impairments. Importantly, as the Canadian health care system shifts towards day surgeries and outpatient settings as opposed to in-hospital care, the development of patient-led strategies to mitigate skeletal muscle disuse atrophy has become increasingly vital.

For most ACLR outpatients, resistance exercise is not feasible in the immediate 2-week post-surgical period, during which the rates of skeletal muscle mass and strength loss are highest. Outside of pharmacology, nutrition represents one alternative strategy to combat skeletal muscle-disuse atrophy during this time. Previous work reported that daily supplementation with EAA prior to and after total knee arthroplasty surgery attenuated skeletal muscle atrophy and enhanced recovery of functional mobility in adults. Similarly, chronic daily supplementation with omega-3 fatty acids reduced declines in quadriceps volume in healthy, young women during single-leg immobilization. This finding complemented previous work in which supplementation with omega-3 fatty acids potentiated muscle protein synthesis rates in response to an hyperaminoacidemic-hyperinsulinemic clamp, but not fasting rates in healthy younger, middle-aged, and older adults, while it additionally improved skeletal muscle strength and power. Together, these data suggest that combined intake of omega-3 fatty acids and EAAs may be an effective strategy to combat skeletal muscle-disuse atrophy, and perhaps loss of skeletal muscle strength, in response to ACLR.

Whilst there is a growing body of literature to promote EAA and omega-3 fatty acids as anabolic stimuli, no work has explored the combined effect of these nutritional strategies in the pathophysiological context of surgery. Nutritional strategies represent an accessible treatment for skeletal muscle disuse atrophy that is independent of patient age, mobility, or current health status, which could prove favourable for surgical outpatients, as well as individuals experiencing periods of prolonged immobilization or bed rest. The future goal of this design is to test efficacy of the combined nutritional strategy of daily omega-3 fatty acid and EAA supplementation to attenuate of skeletal muscle disuse atrophy following elective knee surgery. However, the aim of the present randomized controlled pilot trial is to explore the feasibility of recruitment and retention of adult ACLR outpatients from a single centre across 18 months for a protocol that prescribes combination omega-3 fatty acid and EAA supplementation vs. a calorie- and nitrogen-matched placebo control supplement 4 weeks before and 2 weeks after ACLR surgery. This pilot will also characterize measurements of skeletal muscle volume, strength, and function, and integrated rates of skeletal muscle protein synthesis, as well as report participant adherence to protocols and the incidence of adverse events. The investigators envisage that the data generated from this trial will be used to inform the future large scale randomized controlled trial (RCT) that will examine the effect of the combined nutritional intervention on skeletal muscle volume and functional outcomes in response to ACLR. The results of future work may inform clinical practice and outpatient care guidelines to minimize loss of skeletal muscle mass and strength in response to elective surgery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed anterior cruciate ligament injury requiring reconstruction surgery
* Surgery in Kingston, ON
* Patellar tendon graft, quadriceps tendon graft, or hamstring tendon graft reconstruction procedure

Exclusion Criteria:

* Any muscular, neurological, respiratory, or metabolic disease, subject to investigators' discernment, would negatively affect the subject's ability to comply with the study requirements
* Any form of cancer currently or in the last 5 years
* Bleeding disorders or antiplatelet / anticoagulation therapy
* Currently taking fish oils or within the last 6 months
* Regular consumption (≥ 2x week) of fish oil or oily fish in the last 6 months
* Allergy or sensitivity to fish, shellfish or safflower oils
* Currently taking any form of steroid or within the last 6 months
* Medical inability to attain magnetic resonance imaging scans
* Known irregular responses to physical activity (e.g., shortness of breath, chest pain, dizziness, etc.)
* Surgery scheduled outside of research centre
* Scheduled surgery date < 5 weeks away
* Pregnant or plans to become pregnant within the next 6 months
* Any current illness that impacts ability to participate in protocols

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-10-14 (Actual)

PRIMARY OUTCOMES:
Feasibility of Recruitment and Retention | 18 months and 12 weeks (8 weeks post surgery), respectively.
  Number of participants recruited and retained. Criteria for success is 30 outpatients recruited and at least 22 retained.

SECONDARY OUTCOMES:
Muscle Mass | 0 and 2 weeks
  Change in quadriceps muscle mass measured by magnetic resonance imaging scan.
Muscle Cross-Sectional Area | 0 and 2 weeks
  Change in quadriceps muscle cross sectional area measured by magnetic resonance imaging scan.
Muscle Protein Synthesis | -1 to 0 weeks and 0 to 2 weeks.
  Muscle protein synthesis measured as fractional synthesis rate using combined protocol of skeletal muscle biopsy, stable isotope tracing, cavity ring down spectroscopy with liquid isotope analysis, and gas-chromatography pyrolysis isotope-ratio mass spectrometry.
Skeletal Muscle Phospholipid Composition | -4 and 2 weeks.
  Phospholipid composition will be assessed by gas chromatography.
Erythrocyte Phospholipid Composition | -4 and 2 weeks.
  Phospholipid composition will be assessed by gas chromatography.
Plasma Proteomics | -4, 0 and 2 weeks.
  Change in target signal intensity and protein concentration measured through proteome profiling by aptamer based SOMAscan assay.
Expression of Translational Factors Related to Skeletal Muscle Protein Synthesis | -4, 0 and 2 weeks.
  Activation of translational factors involved in skeletal muscle protein synthesis assessed by western blotting.
Muscle Function | -4 and 8 weeks.
  Stair climb power test performance.
Muscle Strength | -4 and 8 weeks.
  Knee-extensor peak torque measured by dynamometry.
Muscle Power | -4 and 8 weeks.
  Isotonic power measured by dynamometry.

CONTACTS AND LOCATIONS:
Overall Officials: Chris McGlory, PhD, Principal Investigator — Queen's University
Locations (1):
- Queen's University, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nyman DLE, Pufahl CJ, Hickey OGV, Stokes T, Simpson CA, Selinger JC, Mathur S, Janssen I, Giangregorio LM, Bardana DD, McGlory C. Nutritional intervention to enhance recovery after arthroscopic knee surgery in adults: a randomized controlled pilot trial. Pilot Feasibility Stud. 2024 Nov 12;10(1):138. doi: 10.1186/s40814-024-01561-w. PMID 39533408